CLINICAL TRIAL: NCT03346811
Title: Efficiency of Icotinib in Plasma ctDNA EGFR Mutation-positive Patients Diagnosed With Lung Cancer：a Single Arm，Multi-center，Open-label Study
Brief Title: Efficiency of Icotinib in Plasma ctDNA EGFR Mutation-positive Patients Diagnosed With Lung Cancer
Acronym: CHALLENGE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV90
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Plasma EGFR Mutation-positive Lung Cancer
MeSH Terms: interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: icotinib (Experimental): Patients diagnosed with lung cancer with plasma EGFR mutation-positive are arranged to receive icotinib with a dose of 125 mg three times per day, till progressive disease or unaccepted toxicity
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Patients with plasma EGFR mutation-positive are arranged to receive icotinib with a dose of 125 mg three times per day, till progressive disease or unaccepted toxicity
  Other Names: conmana

SUMMARY:
this single arm，open-label，multi-center study is aimed to evaluate the efficiency of icotinib in plasma ctDNA EGFR mutation-positive patients diagnosed with lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of peripheral lung cancer, but the pathological diagnosis is not yet clear.
* Plasma EGFR mutations (EGFR 19del and/or 21L858R) positive (simultaneously detected by Super-ARMS, ddPCR and NGS，any positive).
* unavailable of radical surgery or radical radiotherapy.
* not previously received anticancer therapy like surgery, chemotherapy, radiation therapy, and biotherapy etc.
* Palliative radiotherapy for bone metastases is permitted, but there is no continuous toxicity associated with radiation therapy.
* Age 18-75 years old with performance status of 0 to 3.
* With a measurable disease(longest diameters >=10mm with Spiral computed tomography (CT)) according to RECIST Criteria.None of the lesions treated with radiotherapy could be used as target lesions.
* Adequate hematological, biochemical and organ functions.

Exclusion Criteria:

* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.
* Evidence of interstitial lung diseases
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
* Other situations researchers think not appropriate to enter the group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-18 (Estimated); Primary Completion 2019-05-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 weeks
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | 12 months
  Progression-free survival
DCR | 12 months
  disease control rate
OS | 20 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu J, Liu Z, Bai H, Dong G, Zhong J, Wan R, Zang A, Li X, Li Q, Guo J, Du N, Zhong D, Huang Y, Lv Q, Zhang J, Zhao Y, Gao L, Li L, Zhang C, Zhao J, Li B, Liu Z, Yang Z, Ji D, Wang T, Duan J, Wang Z, Wang J. Evaluation of Clinical Outcomes of Icotinib in Patients With Clinically Diagnosed Advanced Lung Cancer With EGFR-Sensitizing Variants Assessed by Circulating Tumor DNA Testing: A Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2022 Sep 1;8(9):1328-1332. doi: 10.1001/jamaoncol.2022.2719. PMID 35862035